CLINICAL TRIAL: NCT03720548
Title: A Single-Dose and Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3372993 in Healthy Subjects and Patients With Alzheimer's Disease
Brief Title: A Study of LY3372993 in Healthy Participants and Participants With Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17019; J1G-MC-LAKA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3372993 (Part A) (Experimental): LY3372993 administered intravenously (IV) to healthy participants.
  Interventions: Drug: LY3372993
- Placebo (Part A) (Placebo Comparator): Placebo administered IV to healthy participants.
  Interventions: Drug: Placebo
- LY3372993 (Part B) (Experimental): LY3372993 administered IV to participants with AD. Part B was terminated before any participants received treatment.
  Interventions: Drug: LY3372993
- Placebo (Part B) (Placebo Comparator): Placebo administered IV to participants with AD. Part B was terminated before any participants received treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3372993 — Administered IV.
  Arms: LY3372993 (Part A); LY3372993 (Part B)
Drug: Placebo — Administered IV.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3372993 in healthy participants and participants with AD. The study will also investigate how much LY3372993 gets into the bloodstream and test the effects of LY3372993 in participants with AD.

The study has two parts:

* Part A - Healthy participants will receive LY3372993 or placebo. Part A will last up to 17 weeks;
* Part B - Participants with AD will receive LY3372993 or placebo. Part B will last about 317 days.

DETAILED DESCRIPTION:
In April, 2019, Eli Lilly and Company made a business decision to terminate Part B. No participants were enrolled.

ELIGIBILITY:
Inclusion Criteria :

Part A:

* Overtly healthy males or females as determined by medical history and physical examination
* Are between 18 to 45 years old, inclusive
* Male participants agree to use a reliable method of birth control during the study and 3 months following the last dose of the investigational product
* Female participants not of child-bearing potential
* Have a body mass index of 18.0 to 32 kilograms per square meter (kg/m²) inclusive

Part B:

* Present with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or mild-to-moderate AD
* Positive florbetapir scan
* Men or nonfertile women, at least 55 years of age. Nonfertile is defined as hysterectomy and/or bilateral oophorectomy, or amenorrhea for at least 1 year
* Have up to 2 study partners who can provide health information related to the study about the participant. Study partner(s) will provide a separate written informed consent to participate

Exclusion Criteria:

* Have significant abnormalities in brain magnetic resonance imaging (MRI); or have contraindications for MRI
* Have significant allergic reactions to LY3372993, or related compounds, or have significant allergies to humanized monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone
* Have clinically significant neurological or psychological illness, or other illnesses that could affect the study results

Part A:

* Have family history of early onset Alzheimer's Disease (AD)
* Have impaired cognitive function

Part B:

* History of intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, or carotid artery occlusion, or stroke or epilepsy
* Previously dosed in any other study investigating active immunization against amyloid beta (Aβ)
* Previously dosed in any other study investigating passive immunization against Aβ within the last 6 months
* Have current serious or unstable illnesses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 562
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of LY3372993 After a Single Dose | Predose up to Day 85
  PK: AUC of LY3372993 After a Single Dose
PK: Maximum Observed Concentration (Cmax) of LY3372993 After a Single Dose | Predose up to Day 85
  PK: Cmax of LY3372993 After a Single Dose
PK: AUC of LY3372993 at Steady State after Multiple Doses | Week 14 through Week 18
  PK: AUC of LY3372993 at Steady State after Multiple Doses
PK: Cmax of LY3372993 at Steady State After Multiple Doses | Week 14 through Week 18
  PK: Cmax of LY3372993 at Steady State After Multiple Doses
Pharmacodynamics (PD): Change from Baseline in Amyloid Load | Baseline, Week 28
  Amyloid load measured by florbetapir F18 positron emission tomography (PET) scan

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - MD Clinical, Hallandale, Florida
  - BioClinica Inc, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Progressive Medical Research, Port Orange, Florida
  - BioClinica Inc, The Villages, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Carolina Phase 1 Research (Wake M3), Raleigh, North Carolina
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No